CLINICAL TRIAL: NCT00381888
Title: Women's Cancer Center Protocol #45: Prolonged Venous Thromboembolism Prophylaxis With Fondaparinux in Gynecologic Oncology Patients: An Open Label Phase II Trial
Brief Title: Fondaparinux in Preventing Blood Clots in Patients Undergoing Surgery for Gynecologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000503985; UMN-2006LS009 (Other: Clinical Trials Office, University of Minnesota); UMN-0603M82707 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Sarcoma; Thromboembolism; Vaginal Cancer; Vulvar Cancer
Keywords: thromboembolism; cervical cancer; endometrial cancer; ovarian epithelial cancer; ovarian germ cell tumor; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; ovarian stromal cancer; uterine sarcoma; vaginal cancer; vulvar cancer; fallopian tube cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma; Thromboembolism; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Treated with Fondaparinux (Experimental): Patients treated with at least one dose of Fondaparinux (2.5 mg subcutaneous, Days 1-28 by mouth).
  Interventions: Drug: fondaparinux sodium

INTERVENTIONS:
Drug: fondaparinux sodium — Fondaparinux, 2.5 mg subcutaneous, Days 1-28 by mouth.
  Other Names: Artixtra(R)

SUMMARY:
RATIONALE: Fondaparinux may help prevent blood clots from forming in patients who are undergoing surgery for gynecologic cancer.

PURPOSE: This phase II trial is studying how well fondaparinux works in preventing blood clots in patients undergoing surgery for gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of prolonged (4 weeks) fondaparinux sodium administration in venous thromboembolism prophylaxis in patients undergoing gynecologic oncology surgery.

Secondary

* Evaluate the safety of this regimen in these patients (4 weeks).
* Determine the feasibility of this regimen in these patients (4 weeks).

OUTLINE: This is an open-label study.

Beginning after surgery, patients receive fondaparinux sodium subcutaneously once daily on days 1-28 in the absence of disease progression or unacceptable toxicity. Patients undergo duplex ultrasonography of the lower extremities between day 28-35.

ELIGIBILITY:
Inclusion Criteria

* Scheduled to undergo major, open abdominal-pelvic surgery for known or presumed gynecologic malignancy
* Age 18 years or older at the time of signing the consent
* Gynecologic Oncology Group (GOG) performance status of ≤ 2
* Life expectancy of > 3 months
* Patient's weight must be ≥ 50 kg
* Adequate organ function within 28 days of study entry defined as:

  * Hemoglobin ≥ 9.0 g/dL
  * Platelet ≥ 100,000 x 109/L
  * Blood urea nitrogen (BUN) ≤ 30 mg/dL
  * Serum creatinine ≤ 1.5 mg/dL
* Not pregnant as determined by a negative urine or serum pregnancy test within 14 days of study enrollment
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria

* Current treatment with anticoagulants
* Thromboembolism within the previous 6 months
* Bleeding/blood disorders (e.g., thrombocytopenia), gastrointestinal bleeding (e.g., active ulcers), history of stroke within past 3 years, or severe and currently uncontrolled high blood pressure
* Bacterial endocarditis
* Known hypersensitivity to fondaparinux sodium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Crozer-Chester Medical Center, Upland, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Enrolled and Consented: This number includes all patients consented and enrolled in this study.
Period: Overall Study
Arm/Group | Patients Enrolled and Consented
Started | 44
Completed | 27
Not Completed | 17
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 9
Not completed — Had laparoscopic surgery | 2
Not completed — Surgery was cancelled | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients Enrolled and Consented: This number includes all patients that were consented and enrolled in the study and received at least one dose of study drug.
Arm/Group | Patients Enrolled and Consented
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: Years] | 55.7 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Venous Thromboembolism at Week 4
Description: Venous thromboembolism is the formation of a blood clot (thrombus) inside a blood vessel, obstructing the flow of blood through the circulatory system.
Time Frame: Week 4 (Days 28-35)
Population: The number includes those patients who completed the study and are evaluable for this outcome measure.
Measure: Number; unit: Participants
Groups:
- Fondaparinux Patients Who Completed Study: This number includes all patients that completed 4 weeks of the study and were treated with 2.5 mg of Fondaparinux on days 1-28.
Arm/Group | Fondaparinux Patients Who Completed Study
Number analyzed (Participants) | 27
Participants | 0

2. Secondary Outcome: Number of Patients Who Achieved Thromboembolism Prophylaxis at Week 4.
Description: This is a count of patients who did not have a clot (thromboembolism) occur during the 4 weeks of study - attributed to the use of Fondaparinux (study dry). Prophylaxis is a measure taken for the prevention of a disease or condition.
Time Frame: Week 4
Population: These patients completed the study and are considered evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fondaparinux Patients Who Completed Study
Number analyzed (Participants) | 27
Participants | 27

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: 33 of 44 patients received at least one dose of Fondaparinux and therefore have been assessed for toxicity.
Groups:
- All Patients Who Received at Least One Dose of Fondaparinux: This number includes all patients that received one or more doses of study drug. All events were determined to be unrelated to Fondaparinux.
Arm/Group | All Patients Who Received at Least One Dose of Fondaparinux
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Who Received at Least One Dose of Fondaparinux (N=33)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) — Grade 5, death
Colitis (C. difficile) (Infections and infestations) | 1 (1) — Grade 3, severe
Infection/Sepsis (Infections and infestations) | 1 (1) — Grade 5, death
Partial small bowel obstruction (Gastrointestinal disorders) | 1 (1) — Grade 2, moderate
Port-a-cath infection (Infections and infestations) | 1 (1) — Grade 3, severe
Pulmonary embolism, post-op (Vascular disorders) | 1 (1) — Grade 4, life-threatening
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5, death
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) — Grade 4, life threatening
Wound infection (Infections and infestations) | 1 (1) — Grade 2, moderate
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Who Received at Least One Dose of Fondaparinux (N=33)
Anxiety, increased (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 7 (7)
Chills (General disorders) | 1 (1)
Cold sensation, upper thighs & lower abdomen (Nervous system disorders) | 1 (2)
Decreased appetite (anorexia) (Gastrointestinal disorders) | 1 (1)
Dehyration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Emesis (vomiting) (Gastrointestinal disorders) | 4 (4)
Fever (General disorders) | 5 (7)
Heartburn (dyspepsia) (Gastrointestinal disorders) | 1 (1)
Hematoma, retroperitoneal (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (oxygen desaturation) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection, wound (Infections and infestations) | 1 (1)
Lung crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Numbness (paresthesia), upper thighs, lower extremity, abdomen (Nervous system disorders) | 2 (3)
Pain, chest (General disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleeplessness (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Urine output, low (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2)
Vertigo (Nervous system disorders) | 1 (1)
Wound, draining (Skin and subcutaneous tissue disorders) | 3 (3)
Wound, open (Skin and subcutaneous tissue disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No